CLINICAL TRIAL: NCT02154243
Title: An Open Label Trial to Decrease Signs and Symptoms of Orthostatic Hypotension Using Midodrine in Patients With Preserved Cardiac Output (CO) and an Intravenous Fluid Bolus for Patients With Low CO Following Total Hip Arthroplasty
Brief Title: An Open Label Trial to Decrease Signs and Symptoms of Orthostatic Hypotension Using Midodrine or Intravenous Fluid Bolus in Patients Following Total Hip Arthroplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-114
Record Dates: First submitted 2014-05-28; First posted 2014-06-03 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Orthostatic Hypotension
MeSH Terms: conditions — Hypotension, Orthostatic | interventions — Midodrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Midodrine (Experimental): Patients who are diagnosed with orthostatic hypotension at their first physical therapy session and have an SVV<15 will be given oral midodrine, 10 mg, once.
  Interventions: Drug: Midodrine
- Intravenous fluid bolus (Experimental): Patients who are diagnosed with orthostatic hypotension at their first physical therapy session and have an SVV>=15 will be given intravenous fluid bolus, 15 cc/kg, once.
  Interventions: Other: Intravenous fluid bolus
- Control (no intervention) (No Intervention): Patients who are NOT diagnosed with orthostatic hypotension at their first physical therapy session will be given the interventions.

INTERVENTIONS:
Drug: Midodrine — 10 mg, p.o., once, on day of surgery after first physical therapy session
  Other Names: ProAmatine
  Arms: Midodrine
Other: Intravenous fluid bolus — 15 cc/kg, once, on day of surgery after first physical therapy session
  Arms: Intravenous fluid bolus

SUMMARY:
Orthostatic hypotension following total hip arthroplasty is known to limit the ability of patients to perform physical therapy (PT) and increase the length of hospital stay and costs. Our goal is to prospectively study the effects of oral midodrine on the signs and symptoms of orthostatic hypotension in 20 patients and the effects of intravenous fluid on the signs of symptoms of orthostatic hypotension in 10 patients. Midodrine will be administered to patients with suspected low SVV, and an intravenous fluid bolus will be administered to patients with low CO. 120 patients will be consented with a view to studying 30 patients who meet the inclusion criteria for orthostatic hypotension. Patients who receive midodrine or the fluid bolus will undergo hemodynamic measurements at 30 min, 1 hr, 2 hrs, 3 hrs, and 4 hrs post-intervention. All patients will undergo measurements for blood pressure, arterial augmentation index, and heart rate at baseline (pre-op; holding area) and the time of first PT attempt. Patients will be monitored up to post-operative day 3. The working hypothesis is that midodrine or fluid therapy will significantly raise the mean arterial blood pressure (MAP) by 5 mmHg+ and/or cause a significant change in the Orthostatic Hypotension Questionnaire (characterized by a two-point improvement in symptom score).

ELIGIBILITY:
Inclusion Criteria:

* Patients of participating surgeons undergoing unilateral primary total hip arthroplasty
* Ages 18-90
* English-speaking
* If the patients are diagnosed with orthostatic hypotension (fall in SBP of at least 20 mmHg or DBP of at least 10 mmHg within 3 min of assuming a sitting/standing position)

Exclusion Criteria:

* Body mass index > 40
* Low ejection fraction (<50%)
* Clinical diagnosis of congestive heart failure
* Aortic insufficiency characterized as greater than moderate
* Severe uncontrolled hypertension
* Symptomatic bradycardia (HR < 50 bpm and symptoms)
* Creatinine > 1.2 mg/dl
* Hepatic insufficiency
* Severe respiratory disease in which supplemental oxygen is required
* History of severe urinary retention
* Use of MAO inhibitors
* Severe supine hypertension (SBP >= 150 mmHg or DBP >= 90 mmHg)
* History of visual problems and using fludrocortisone acetate
* Contraindication for repeated BP measurements
* Revision THA and additional procedures
* Clonidine use

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Midodrine | Intravenous Fluid Bolus | Control (no Intervention)
Started | 5 | 4 | 4
Completed | 5 | 4 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Midodrine | Intravenous Fluid Bolus | Control (no Intervention) | Total
Number analyzed (Participants) | 5 | 4 | 4 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (11.3) | 55.7 (11.2) | 57.7 (11.2) | 55.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 7
  Male | 2 | 2 | 2 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Orthostatic Hypotension Questionnaire Score
Time Frame: From baseline assessment to post-intervention (30 min, 1 hr, 2 hrs, 3 hrs, 4 hrs)
Population: DATA WAS NOT COLLECTED. STUDY TERMINATED EARLY.
Arm/Group | Midodrine | Intravenous Fluid Bolus | Control (no Intervention)
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

2. Secondary Outcome: Length of Stay
Time Frame: Length of the hospital stay (average of 4 days)
Population: DATA WAS NOT COLLECTED. STUDY TERMINATED EARLY.
Arm/Group | Midodrine | Intravenous Fluid Bolus | Control (no Intervention)
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Midodrine | Intravenous Fluid Bolus | Control (no Intervention)
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes